CLINICAL TRIAL: NCT01065987
Title: Randomized, 2-way Crossover, Bioequivalence Study of Tizanidine Hydrochloride 4mg Tablets and Zanaflex® 4mg Tablets Administered As 1 x 4mg Tablet in Healthy Adult Subjects Under Fed Conditions
Brief Title: Bioequivalence Study of Tizanidine HCl 4mg Tablets of Dr.Reddy's Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Assistant Manager, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 01221
Record Dates: First submitted 2010-02-08; First posted 2010-02-10 (Estimated); Last update posted 2010-02-10 (Estimated); Status verified 2010-02

CONDITIONS: Healthy
MeSH Terms: interventions — tizanidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tizanidine HCl 4 mg (Experimental): Tizanidine HCl Tablets 4 mg, Dr.Reddy's Laboratories Limited
  Interventions: Drug: Tizanidine
- Zanaflex (Active Comparator): Zanaflex 4 mg Tablets
  Interventions: Drug: Tizanidine

INTERVENTIONS:
Drug: Tizanidine — Tizanidine HCl Tablets 4 mg
  Other Names: Zanaflex 4 mg

SUMMARY:
The purpose of this bioequivalence study is to compare the test tizanidine Hydrochloride 4mg tablets of Dr.Reddys Laboratories Limited with reference zanaflex® 4mg tablets of Elan in healthy adult subjects under fed conditions.

DETAILED DESCRIPTION:
Randomized, 2-way crossover, bioequivalence study of tizanidine Hydrochloride 4mg tablets and zanaflex® 4mg tablets administered As 1 x 4mg tablet in healthy adult subjects under fed conditions

ELIGIBILITY:
Inclusion Criteria:

Subjects enrolled in this study will be members of the community at large. The recruitment advertisements may be done using different media (e.g. radio, newspaper, Anapharm Inc.

Web site). Subjects must meet all of the following criteria in order to be included in the study:

* Subjects will be females and/or males, smokers or non-smokers, 18 years of age and older.
* Female subjects will be post-menopausal or surgically sterilized.

  * Post-menopausal status is defined as absence of menses for the past 12 months.
  * Sterile status is defined as hysterectomy, bilateral oophorectomy or tubal ligation at least 6 months ago.

Exclusion Criteria:

Subjects to whom any of the following applies will be excluded from the study:

* Clinically significant abnormalities found during medical screening.
* Clinically significant surgery within 4 weeks prior to the administration of the study medication.

Clinically significant illnesses within 4 weeks of the administration of study medication.

* History of neuromuscular disease.
* Abnormal laboratory tests judged clinically significant.
* ECG abnormalities (clinically significant) or vital sign abnormalities (systolic blood pressure lower than 100 or over 140 mmHg, or diastolic blood pressure lower than 70 or over 90; or heart rate less than 60 bpm) at screening.
* Subjects with BMI ≥ 30.0.
* History of allergic reactions to tizanidine hydrochloride.
* Any food allergies, intolerances, restrictions, or special diet which in the opinion of the medical sub investigator, contraindicates the subject's participation in this study.
* Positive urine drug screen at screening.
* Positive testing for hepatitis B, hepatitis C or HN at screening.
* Positive urine pregnancy test at screening.
* Donation of plasma (500 mL) within 7 days or donation or significant loss of whole blood (500 mL) within 56 days prior to administration of the study medication.
* History of significant alcohol abuse within six months of the screening visit or any indication of the regular use of more than two units of alcohol per day (l Unit = 150 mL of wine or 360 mL of beer or 45 mL of alcohol 40%).
* History of drug abuse or use of illegal drugs: use of soft drugs (such as marijuana, pot) within 3 months of the screening visit or hard drugs (such as cocaine, phencyclidine (PCP) and crack) within 1 year of the screening visit.
* Subjects who have taken prescription medication within 14 days prior to administration of study medication or over-the-counter products within 7 days prior to administration of study medication, except for topical products without systemic absorption.
* Smoking more than 25 cigarettes per day.
* Use of any drugs known to induce or inhibit hepatic drug metabolism (examples of inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, rifampin/rifabutin; examples of inhibitors: antidepressants, cimetidine, diltiazem, erythromycin, ketoconazole, MAO inhibitors, neuroleptics, verapamil, quinidine), use of an investigational drug or participation in an investigational study within 30 days prior to administration of the study medication.
* Any reason which, in the opinion of the medical sub investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2001-09; Primary Completion 2001-09 (Actual); Study Completion 2001-11 (Actual)

PRIMARY OUTCOMES:
Bioequivalence study of Tizanidine HCl Tablets 4 mg of Dr.Reddy's Laboratories Limited under Fed Conditions | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Girard, M.D, Principal Investigator — Anapharm
Locations (1):
- Anapharm Inc., Sainte-Foy (Quebec), Canada